CLINICAL TRIAL: NCT01952951
Title: A Randomized Phase II Trial of Preoperative Chemoradiation (Preop CRT) Followed by CapOx (Capecitabine Plus Oxaliplatin) Versus Preop CRT Alone for Locally Advanced Rectal Cancer (LARC)
Brief Title: Preoperative Chemoradiation Followed by Chemotherapy for Locally Advanced Rectal Cancer
Acronym: PREPARE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Sun Young Kim, MD, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCSG CO14-03
Record Dates: First submitted 2013-09-11; First posted 2013-09-30 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Rectal Neoplasms; Adenocarcinoma
Keywords: rectal neoplasms; radiotherapy; Antineoplastic Agents
MeSH Terms: conditions — Rectal Neoplasms; Adenocarcinoma | interventions — XELOX; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- chemoradiation followed by CapOx (Experimental): preoperative chemoradiation 50.4Gy with capecitabine or 5-fluorouracil/leucovorin (pelvic radiation capecitabine 5-fluorouracil) followed by 2 cycles of chemotherapy (Capecitabine Oxaliplatin - CapOx) and surgery (total mesorectal excision)
  Interventions: Drug: Capecitabine Oxaliplatin; Radiation: pelvic radiation capecitabine 5-fluorouracil
- chemoradiation (Active Comparator): preoperative chemoradiation 50.4Gy with capecitabine or 5-fluorouracil/leucovorin (pelvic radiation capecitabine 5-fluorouracil) followed by rest for 8 weeks and surgery (total mesorectal excision)
  Interventions: Radiation: pelvic radiation capecitabine 5-fluorouracil

INTERVENTIONS:
Drug: Capecitabine Oxaliplatin — after completion of chemoradiation, two cycles of capecitabine (850mg/m2 twice daily from D1 evening to D15 morning) and oxaliplatin (100mg/m2 on D1) will be administered every 3 weeks.
  Other Names: Xeloda; Oxalitin
  Arms: chemoradiation followed by CapOx
Radiation: pelvic radiation capecitabine 5-fluorouracil — 50.4Gy of pelvic radiation with capecitabine or 5-fluorouracil
  Other Names: preoperative chemoradiation; xeloda

SUMMARY:
The current standard treatment of locally advanced rectal cancer (clinical stage II or III) is preoperative radiation with chemotherapy (CRT) followed by surgery. But this approach can be suboptimal for patients with high risk features (more deeply-seated tumor or many regional lymph nodes involved)that are associated with recurrence. This study test a hypothesis that CRT followed by chemotherapy before surgery can improve efficacy of preoperative treatment.

DETAILED DESCRIPTION:
Downstaging rate with CRT using fluoropyrimidine monotherapy is usually 30-40%.In MRI-defined high-risk patients, downstaging rate with conventional fluoropyrimidine-based monotherapy with radiation has not been shown. We assume that the downstaging rate of chemoradiation arm (control arm) would be 30%, and that addition of CapOx after CRT (experimental arm) may increase downstaging rate 30% to 50%. A sample size of 52 patients per group is needed have 85% power to detect downstaging rate = 50% as compared to 30% with type I error rate of 15%. We will perform one interim futility analysis when half of the patients are recruited and evaluated for the primary endpoint. O'Brien-Fleming boundary will be considered. Therefore, when 26 patients per arm are evaluated, the interim futility analysis will be performed, and when the Z score at the interim is less than -0.09192 (one-sided p-value greater than 0.5366192), the study will be stopped for futility. Considering 5% follow-up loss, a sample size of 55 per arm (a total of 110 patients) will be studied.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed adenocarcinoma of the rectum
* distal margin of tumor located from 0 to 12 cm from anal verge measured by digital rectal examination
* high risk clinical stage II or III in MRI (satisfying at least one of the followings)

  * circumferential resection margin < 1 mm involved
  * low-lying tumor below anal verge 3 cm
  * T3 > 5 mm extramural spread
  * T4 (involving surrounding structures or peritoneum)
  * cN2 (4 or more mixed signal intensity or irregularly bordered node or tumor deposit)
* age 20 years or more
* ECOG (Eastern Cooperative Oncology Group) performance status 0-2
* No prior chemotherapy, radiotherapy to pelvis
* Adequate bone marrow function
* Adequate renal function
* Adequate hepatic function
* patients must sign the informed consent indicating that they were aware of the investigational nature of the study in keeping with the policy of the hospital

Exclusion Criteria:

* malignant disease of the rectum other than adenocarcinoma or arisen from chronic inflammatory bowel disease
* any unresected synchronous colon cancer
* any distant metastases
* intestinal obstruction or impending obstruction, but decompressing colostomy is permitted
* any previous or concurrent malignancy withih 5 years other than non-melanoma skin cancer / in situ cancer of uterine cervix / early gastric cancer / thyroid cancer of low risk
* any other morbidity or situation with relative contraindication for chemoradiotherapy
* patients with history of significant gastric or small bowel resection, or malabsorption syndrome, or other lack of integrity of the upper gastrointestinal tract that may compromise the absorption of capecitabine
* pregnant or lactating women or patients of childbearing potential not predicting adequate contraception

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-06; Primary Completion 2017-09 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
downstaging rate | expected average of 15 weeks after start of study treatment
  downstaging rate is defined as the proportion of patients with ypStage (pathologic stage after preoperative treatment) 0 or I (from pathologic findings after preoperative treatment and surgery) out of all patients who were assigned to each arm.

SECONDARY OUTCOMES:
pathologic response | expected average of 15 weeks after start of study treatment
  pathologic response is assessed by Dworak's grading system from postoperative specimen.
radiologic response rate | expected average of 14 weeks after start of study treatment
  radiologic response will be assessed according to RECIST (Response Evaluation Criteria in Solid Tumors) guideline 1.1
toxicity profile | expected average of 35 weeks after start of study treatment
  Toxicities or any adverse events during study treatment, surgery and follow-up period will be assessed according to NCI CTCAE (Common Terminology Criteria for Adverse Events) version 4.0
pattern of failure | 3 years after surgery
  if any recurrent lesion is noticed, anatomic sites of recurrent lesions and the date and the name of exam or imaging study (physical exam, CT or MRI…) will be recorded in case report form.
local control rate | 3 years after surgery
  Local recurrence is defined as tumor recurrence confined in radiation field (pelvic cavity). Cumulative incidence of local recurrence will be suggested.
relapse-free survival | 3 years after surgery
  Time from date of operation to date of recurrence of disease or deaths due to recurrence or progression of disease.
Disease-free survival | 3 years after surgery
  time from date of operation to date of recurrence of disease, a new occurrence of secondary colorectal cancer, a new occurrence of other malignancy, or deaths from any cause.
overall survival | 3 years after surgery
  time from date of operation to date of death due to any cause.
quality of life | before study treatment, 7 weeks after completion of chemoradiation, and at 4 weeks after surgery
  quality of life will be measured with FACT-C

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young Kim, MD, Study Chair — Asan Medical Center
Locations (7):
- South Korea (7):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Anyang
  - Gangneung Asan Hospital, Gangneung
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim SY, Joo J, Kim TW, Hong YS, Kim JE, Hwang IG, Kim BG, Lee KW, Kim JW, Oh HS, Ahn JB, Zang DY, Kim DY, Oh JH, Baek JY. A Randomized Phase 2 Trial of Consolidation Chemotherapy After Preoperative Chemoradiation Therapy Versus Chemoradiation Therapy Alone for Locally Advanced Rectal Cancer: KCSG CO 14-03. Int J Radiat Oncol Biol Phys. 2018 Jul 15;101(4):889-899. doi: 10.1016/j.ijrobp.2018.04.013. Epub 2018 Apr 12. PMID 29976501